CLINICAL TRIAL: NCT04729660
Title: Efficacy of Kinesio Taping on Mutational Falsetto: A Randomized, Double-blind, Sham-controlled Clinical Trial
Brief Title: Efficacy of Kinesio Taping on Mutational Falsetto
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization (Other)
Responsible Party: Principal Investigator, Yavuz Atar, Associate Professor, M.D., Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 310
Record Dates: First submitted 2021-01-21; First posted 2021-01-28 (Actual); Last update posted 2021-02-04 (Actual); Status verified 2021-02

CONDITIONS: Mutational Falsetto; Dysphonia
Keywords: kinesio taping; mutational falsetto; therapy; dysphonia
MeSH Terms: conditions — Dysphonia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Study group (Active Comparator): Evaluate of the Kinesio tex gold tape that applied to anterior neck localised.
  Interventions: Device: Kinesio Tex Gold
- Sham group (Sham Comparator): Evaluate of the Kinesio tex gold tape that applied to different neck localised as no-stretched.
  Interventions: Device: Kinesio Tex Gold

INTERVENTIONS:
Device: Kinesio Tex Gold — The Kinesio Tex Gold is a kinesio tape that had been certified and patented.

SUMMARY:
This study aimed to assess of efficacy of the kinesio-taping on male patients suffering from mutational falsetto

DETAILED DESCRIPTION:
Mutational falsetto is a functional voice disorder involving a failure to transition from the high-pitched voice of childhood to the lower-pitch ed voice of adolescence and adulthood. In the recent years, kinesio taping has begun to be employed for treating dysphonia patients. We hypothesized that, because the kinesio taping relaxes the suprahyoid muscles and pushes the larynx backward, it could also be used as a therapy of mutational falsetto. This study aimed to assess of efficacy of the kinesio taping on male patients suffering from mutational falsetto.

ELIGIBILITY:
Inclusion Criteria:

* Patients suffered from Mutational falsetto
* Patients who were accept to consent form
* Patients who have not open wound on neck

Exclusion Criteria:

* Having mental disorders or major physiatric disorders
* Cognitive limitations
* Contact dermatitis
* history of smoking
* Asthma, chronic pulmonary diseases
* history of allergic reactions against to medical tape applied
* having an other organic vocal disorders
* advanced hearing loss
* Out of BMI<18.5 or 30<BMI
* Out of age 16-60 years old patients who were not accept to consent form.

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — The males show more commonly that findings of mutational falsetto.
Enrollment: 30 (Actual)
Dates: Start 2020-07-31 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2021-01-31 (Actual)

PRIMARY OUTCOMES:
The outcomes of voice handicap index - 10 | Baseline
  It was assessed by voice handicap index - 10 that a self questionnaire in mutational falsetto patients. The minimum score is 0 and maximum score is 4 per question. The high scores were worst low scores were good.
The outcomes of voice handicap index - 10 | 2 weeks
  It was assessed by voice handicap index - 10 that a self questionnaire in mutational falsetto patients. The minimum score is 0 and maximum score is 4 per question. The high scores were worst low scores were good.
The outcomes of Grade-Roughness-Breathiness-Asthenia-Strain scale | Baseline
  It was assessed by Grade-Roughness-Breathiness-Asthenia-Strain scale that a scale in mutational falsetto patients. The minimum score is 0 and maximum score is 3 per category. The high scores were worst low scores were good.
The outcomes of Grade-Roughness-Breathiness-Asthenia-Strain scale | 2 weeks
  It was assessed by Grade-Roughness-Breathiness-Asthenia-Strain scale that a scale in mutational falsetto patients. The minimum score is 0 and maximum score is 3 per category. The high scores were worst low scores were good.
The outcomes of fundamental frequency | Baseline
  It was analyzed with noise harmonic ratio, jitter and shimmer that were calculated by computer software. Typical average values for the frequencies are 120 Hz for men and 210 Hz for women. The lower frequencies show masculine voice. The higher frequencies show feminine voices.
The outcomes of fundamental frequency | 2 weeks
  It was analyzed with noise harmonic ratio, jitter and shimmer that were calculated by computer software. Typical average values for the frequencies are 120 Hz for men and 210 Hz for women. The lower frequencies show masculine voice. The higher frequencies show feminine voices.
The outcomes of maximum phonation times | Baseline
  The subjects tried to say the vowel "a'" for as long as they could than it was assessed as seconds.
  Typical average values for the maximum phonation times are between 15-30 seconds. The higher times show healthy phonation.
The outcomes of maximum phonation times | 2 weeks
  The subjects tried to say the vowel "a'" for as long as they could than it was assessed as seconds.
  Typical average values for the maximum phonation times are between 15-30 seconds. The higher times show healthy phonation.

SECONDARY OUTCOMES:
Mean of demographic | Baseline
  Age, gender, history of smoke, history of morbidities, history of treatments, diagnosis, were noted

CONTACTS AND LOCATIONS:
Overall Officials: Yavuz Atar, Asso Prof,MD, Study Chair — University of Health Sciences, Prof Dr Cemil Tascioglu City Hospital
Locations (1):
- Prof Dr Cemil Tascioglu City Hospital, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Background] Salturk Z, Doganay T, Ustun O, Tutar B, Akgun MF, Uyar Y. Efficacy of Low Mandible Maneuver on Mutational Falsetto. Folia Phoniatr Logop. 2021;73(5):442-448. doi: 10.1159/000506631. Epub 2020 Mar 27. PMID 32222704
- [Background] Mezzedimi C, Spinosi M, Mannino V, Ferretti F, Al-Balas H. Kinesio Taping Application in Dysphonic Singers. J Voice. 2020 May;34(3):487.e11-487.e20. doi: 10.1016/j.jvoice.2018.11.001. Epub 2018 Dec 6. PMID 30528384